CLINICAL TRIAL: NCT05336396
Title: Impact of Brief Motivational Interviewing on Periodontal Clinical Outcomes: a 3-year Post-trial Follow-up
Acronym: BMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Principal Investigator, Michelle Arnett, Assistant Professor, University of Minnesota
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DENT-2022-30805
Record Dates: First submitted 2022-04-12; First posted 2022-04-20 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Periodontal Diseases; Plaque Score; Bleeding on Probing; Gingival Index
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI (Experimental)
  Interventions: Other: BMI
- Traditional Oral Hygiene Instruction (No Intervention)

INTERVENTIONS:
Other: BMI — Longitudinal data will be collected to determine the effectiveness of BMI compared to traditional OHI to maintain and improve periodontal health.
  Arms: BMI

SUMMARY:
The objective is a 3-year follow-up clinical trial to evaluate longitudinal indicators of periodontal disease (plaque score, bleeding on probing (BOP), and gingival index (GI)) in 58 participants who completed NCT03571958. These participants were randomized to a brief motivational (BMI) test group or a traditional oral hygiene instruction (OHI) group for a 1-year clinical trial from 2018-2020.

In addition, analysis of retrospective data to determine health topics that emerge from the behavior change strategy of BMI compared to traditional OHI by transcription of audio recordings from 2018-2020.

ELIGIBILITY:
Inclusion Criteria:

° Completed all study visits of STUDY00003697 (NCT03571958)

Exclusion Criteria:

* Current smoker or quit smoking within the last year
* Pregnant, planning to become pregnant, or unsure of pregnancy status (self-reported)
* Uncontrolled diabetes (HbA1C > 7)
* Medical conditions that may influence the outcome of the study (neurologic or psychiatric disorders, systemic infections, cancer, and/or HIV/AIDS)
* Current use of oral bisphosphonates
* History of IV bisphosphonates
* Require pre-medication or on long-term antibiotics
* Current orthodontic treatment or planning to begin orthodontic treatment during the study
* Unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2023-03-25 (Actual); Study Completion 2023-03-25 (Actual)

PRIMARY OUTCOMES:
Plaque score | Recorded one time 2 years +/- 8 months
  Excellent hygiene: 0-20%, Good hygiene: 21-40%, Fair hygiene: 41-60%, Poor hygiene: 61-100%
Bleeding on probing | Recorded one time 2 years +/- 8 months
  Presence of bleeding (yes) or absent of bleeding (no)
Gingival index | Recorded one time 2 years +/- 8 months
  0= normal gingiva, 1=mild inflammation (no BOP), 2=moderate inflammation (BOP), 3=severe inflammation (spontaneous bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Arnett, Principal Investigator — University of Minnesota
Locations (1):
- School of Dentistry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No